CLINICAL TRIAL: NCT04806217
Title: Nature of the Link Between Executive Functions and Theory of Mind in Multiple Sclerosis
Acronym: TDE-SEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P00109
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Theory of Mind; Nonverbal false belief task; Cognitive functions; Inhibition and inference abilities
MeSH Terms: conditions — Multiple Sclerosis; Inhibition, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ¨Patients with multiple sclerosis (Experimental): Patients :
  * With multiple sclerosis
  * Aged of 18 and over
  * Recruited during their consultation in the adult outpatient unit or neurological unit or during a hospitalization.
  Interventions: Other: Theory of Mind

INTERVENTIONS:
Other: Theory of Mind — Patients will be submitted to different neuropsychological tests used in routine and the non-verbal false belief task through in the Theory of Mind

SUMMARY:
The purpose of this study is to explore inhibition and inference abilities in The Theory of Mind skills in multiple sclerosis patients using the Theory of Mind task.

DETAILED DESCRIPTION:
Multiple sclerosis is an autoimmune inflammatory disease of the central nervous system. It can cause lesions responsible for motor, ocular, sensory and cognitive symptoms.

The Theory of Mind and the primary facial emotions recognition (anger, joy, fear, surprise, sadness, disgust) are two processes of social cognition that play a role in the social interactions and social reasoning. The Theory of Mind is defined by the ability to understand the other person including thoughts, beliefs and desires that are unique and that may be different from our own.

In multiple sclerosis, difficulties in social cognition are associated with cognitive disorders, (even if the link with a deficit in executive functions remains debated). Indeed, when attributing a mental state to another person is needed,it is mandatory to put ourselves in the other person's place to adopt another perspective. Thus, several executive functions are required: working memory to maintain and manipulate several perspectives, flexibility to switch from one perspective to another one, and finally the inhibition of our own perspective to adopt the other's point of view.

The Theory of Mind's assessment uses nonverbal false belief task which assesses the ability to inhibit its own perspective to infer the mental state of another and the ability to change its perspective to adopt another's.

Thus, the purpose of this study is to explore inhibition and inference abilities in The Theory of Mind skills in multiple sclerosis patients using the Theory of Mind task.

ELIGIBILITY:
Inclusion Criteria:

People :

* With multiple sclerosis
* Age ≥ 18 years old
* Not objecting to the use of their data

Exclusion Criteria:

* Any associated neurological pathology or severe or chronic somatic disease (cancer)
* Visual and/or auditory disorders that do not allow for test taking
* Uncontrolled major psychiatric disorders
* Recent treatment with corticosteroids (less than 4 weeks before the evaluation)
* Patients under guardianship, curatorship or safeguard of justice
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of correct answers to the "unknown reality" false belief tasks | Day 0
  The number of correct answers to the "unknown reality" false belief tasks out of 12 tests will allow to obtain a mental state inference score
Number of correct answers to the "known reality" false belief tasks | Day 0
  The number of correct answers to the "known reality" false belief tasks out of 12 tests will allow to obtain a score for inhibition of its own perspective

SECONDARY OUTCOMES:
California Verbal Learning Test (CVLT) | Day 0
  Verbal episodic memory abilities will be measured through the Learning test of a 16 words list belonging to 4 distinct semantic categories (flowers, fish, clothes, fruit). The list is presented 5 times to the patient who must remember it immediately after each presentation, after the presentation of a second interfering list and after a 20-minute delay. A main score is extracted.
Brief Visuo-spatial Memory Test (BVMT) | Day 0
  Learning test in episodic visuo-spatial memory of 6 simple geometrical drawings. This test presents 3 phases during which the sheet containing the 6 drawings is presented to the participant for 10 seconds, followed by an immediate recall phase (free hand reproduction of the drawings). A delayed recall phase (at 7 minutes) and a delayed recognition phase (among 12 distractors) is also proposed. A main score is extracted.
Symbol Digit Modalities Test (SDMT) | Day 0
  Coding test in which the patient has 90 seconds to state orally the correspondence of numbers (from 1 to 9) to 9 different symbols (matched according to a matching standard). The correct answers number is measured.
Stroop test | Day 0
  The Stroop test is used to evaluate executive functions, especially inhibition abilities and sensitivity to interference. This test offers 3 situations in which performance is measured by the time taken by the patient for each situation and the number of uncorrected errors.
Trail Making test | Day 0
  The Trail Making Test is used to evaluate executive functions especially the cognitive flexibility abilities. The subject's performance is evaluated by the time taken by the subject, the total number of errors and the number of perseveration errors.
Verbal fluency test | Day 0
  The verbal fluency test evaluates executive functions, and more specifically the spontaneous flexibility's abilities. The performance is evaluated by the number of different words cited.
Verbal fluency test | Day 0
  The participant in a given time, evokes (orally or in writing) the greatest number of words according to a given instruction, generally according to a semantic or phonemic categorization. A verbal fluency test measures the participant's ease in producing meaningful speech, both qualitatively and quantitatively
Beck Depression Inventory (BDI) | Day 0
  The Beck Depression Inventory is used to assess depressive disorders. It is a 13-items self-questionnaire rated from 0 (no problem) to 3 (maximum severity of this symptom). The depression's severity is assessed by classifying the total score into 3 levels of intensity: <3: Normal; 3-8: Borderline; >8: Depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lenne, Principal Investigator — Hôpital Saint Vincent de Paul, Lille

IPD SHARING:
Plan to Share IPD: No